CLINICAL TRIAL: NCT06625710
Title: A Randomized, Double-blind, Placebo Controlled, Dose-escalation Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics After Single and Multiple Administration of GV1001 in Healthy Subjects
Brief Title: Evaluation of the Safety, Tolerability and PK Characteristics of GV1001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: GV1001-PK-CL1-013
Record Dates: First submitted 2024-09-24; First posted 2024-10-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Neuro-Degenerative Disease
Keywords: Pharmacokinetic Characeristics
MeSH Terms: interventions — GV1001 peptide; Saline Solution

STUDY DESIGN:
Intervention Model Description: There are two sequential arms plus one extra cohort:
  Part A: 2.24 mg and 4.48 mg Part B: 0.56 mg, 1.12 mg, 2.24 mg, and 4.48 mg Extra cohort: 1.12 mg, 8 Caucasian, after completion of dose group 1.12 in Part B.
  All dose groups will recruit participants at a ratio of 6:2 for the study drug to placebo.
  All dose escalation between dose groups and from Part A to Part B will be determined by the SRC's review and must be carried out sequentially.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A-1 (Experimental): GV1001 2.24 mg SAD or Placebo
  Interventions: Drug: GV1001; Drug: Placebo
- Part A-2 (Experimental): GV1001 4.48 mg SAD or Placebo
  Interventions: Drug: GV1001; Drug: Placebo
- Part B-1 (Experimental): Part B-1: GV1001 0.56 mg MAD (6 treatments for 2 weeks)
  Interventions: Drug: GV1001; Drug: Placebo
- Part B-2 (Experimental): GV1001 1.12 mg MAD or Placebo (6 treatments for 2 weeks )
  Interventions: Drug: GV1001; Drug: Placebo
- Part B-3 (Experimental): GV1001 2.24 mg MAD or Placebo (6 treatments for 2 weeks)
  Interventions: Drug: GV1001; Drug: Placebo
- Part B-4 (Experimental): GV1001 4.48 mg MAD or Placebo (6 treatments for 2 weeks)
  Interventions: Drug: GV1001; Drug: Placebo
- Extra Cohort (Experimental): GV1001 1.12 mg MAD or Placebo (6 treatments for 2 weeks ), Caucasian Only
  Interventions: Drug: GV1001; Drug: Placebo

INTERVENTIONS:
Drug: GV1001 — Lyophilized peptide from hTERT
  Other Names: Tertomotide
Drug: Placebo — 0.9 % Normal Saline
  Other Names: Normal saline

SUMMARY:
The goal of this clinical trial is to assess the the safety, tolerability and pharmacokinetic characteristics after single and multiple administration of GV1001 in healthy subjects. The main questions it aims to answer are:

Safety and Tolerability of GV1001 in different dose scheme, and PK Characteristics of GV1001 in differenct dose scheme

Part A: single dose, 8 days clinical trial participation including one 3-day hospitalization

Part B & Extra Cohort: Multiple dose, 42 days clinical trial participation (12 days treatment + 30 days safety follow-up) including two times of 3-day hospitalization.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, dose-escalation phase 1 clinical trial to evaluate the safety, tolerability and pharmacokinetic characteristics after single and multiple administration of GV1001 in healthy subjects.

The study is divided into Part A and Part B. Part A focuses on assessing the safety, tolerability, and pharmacokinetic characteristics following a single subcutaneous (SC) administration of the GV1001. Part B aims to evaluate the safety, tolerability and pharmacokinetic characteristics following multiple administrations of GV1001. The dose escalation between each dosage group and the transition from Part A to Part B will be determined by the Safety Review Committee (SRC), based on the safety and tolerability data obtained from the previous dose and Part A. The Safety Review Committee (SRC) is an independent committee that reviews safety data while maintaining blind.

An Extra Cohort to assess the safety, tolerability, and pharmacokinetic characteristics of GV1001 in Caucasians can be implemented sequentially after the safety review by the SRC for the 1.12 mg dose group in Part B has been completed.

Screening tests will be conducted within 4 weeks of IP administration to select participants deemed suitable for the clinical trial. In this process, informed consent will be obtained, and a screening number will be assigned to the participants.

Part A - Single Dose Participants deemed suitable for Part A will be admitted on Day -1. On Day 1 at 9 AM, after fasting, they will receive a single SC administration of GV1001 or a placebo. Following this, they will complete the scheduled assessments of the safety, tolerability and pharmacokinetic characteristics and be discharged on Day 3. An end-of-study visit will take place on Day 8 as an outpatient appointment. Dose escalation to the next dose group within Part A will be determined by the SRC's review.

Part B - Multiple Dose Participants deemed suitable for Part B will be admitted on Day -1. On Day 1 at 9 AM, after fasting, participants will receive a single SC administration of GV1001 or a placebo. Following this, they will complete the scheduled assessments of the safety, tolerability and pharmacokinetic characteristics and be discharged on Day 2. Subsequently, participants will receive subcutaneous administrations of GV1001 or placebo in a fasting state during four outpatient visits. At Day 11, participants will be admitted and will complete the scheduled assessments of the safety, tolerability, pharmacokinetic characteristics and the last administration of GV1001 (Day 12). Participants will be discharged on Day 13, and the end of study visit will take place on Day 42, which is 30 days after the last administration. Dose escalation to the next dose group within Part B will be determined by the SRC's review.

The total target number of participants is 56. In Part A, 16 participants will be recruited in two dose groups (2.24 mg and 4.48 mg), while in Part B, 32 participants will be recruited across four dose groups (0.56 mg, 1.12 mg, 2.24 mg, and 4.48 mg). An additional cohort consisting of 8 Caucasian participants is planned, which will be recruited after the completion of the 1.12 mg dose group in Part B. All dose groups will recruit participants at a ratio of 6:2 for the study drug to placebo. All dose escalation between dose groups and from Part A to Part B will be determined by the SRC's review and must be carried out sequentially.

ELIGIBILITY:
Inclusion Criteria:

1. is healthy adults aged between 19 and 50 years at the time of screening. In Part B, only male participants will be included.
2. [Extra Cohort Only] is healthy Caucasian aged between 19 and 50 years at the time of screening.
3. weigh between 50 kg and 90 kg and have a body mass index (BMI) of 18.0 to 27.0.
4. has no skin diseases or skin damage (including scars and tattoos) at the administration site and should not have any medical history that could affect pharmacokinetics (PK)

Exclusion Criteria:

1. has clinically significant or history of liver, kidney, nervous system, respiratory system, endocrine, blood, tumor, cardiovascular, or mental disorders (such as mood disorders, obsessive-compulsive disorder, etc.);
2. has a history of clinically significant hypersensitivity reactions;
3. who showed the following results during the screening test:

   * positive serum test results (Hepatitis B, C test, Human Immunodeficiency Virus (HIV), Syphilis test);
   * [Part B only] testosterone levels outside the normal range (2.67-10.12 ng/ml);
   * [Part B only] Leutinizing hormone (LH) outside the normal range (1.0 - 5.3 mlU/ml); [Part B only] Follicular stimulating hormone (FSH) outside the normal range (1.3 - 8.1 mlU/ml)
4. has a history of substance abuse or those who tested positive for illicit drugs in a urine drug screening.
5. who have taken any prescription medications within 2 weeks prior to the planned first administration, or any over-the-counter (OTC) medications or health supplements within 1 week;
6. who have taken barbiturate-inducing or inhibiting drugs within 1 month prior to the planned first administration;
7. who have participated in another clinical trial or a bioequivalence study within the past 6 months;
8. who have donated whole blood within the past 2 months, or have donated blood components within the past month, or have received a transfusion within the past month prior to planned first administration;
9. who engage in continuous alcohol consumption (over 21 units/week = 10g of pure alcohol) or are unable to abstain from alcohol from 3 days prior to the expected first dosing until the last visit.
10. who are unable to abstain from consuming grapefruit-containing foods or caffeine-containing foods from 3 days prior to the planned first administration of the investigational product (IP) until the post study visit (PSV);
11. who have smoked more than 10 cigarettes per day in the past 3 months, or who cannot abstain from smoking during the clinical trial;
12. who do not use medically acceptable methods of contraception during the clinical trial period;
13. pregnant or breastfeeding women.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Part B and Extra Cohort only recruit healthy male volunteers
Enrollment: 59 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of GV1001 | 6 weeks
  To evaluate the safety and tolerability of GV1001 in healthy adults during both single and multiple administrations in different dose scheme.
  1. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
  2. Number of participants with treatment-related 12-lead ECG abnormality
  3. Number of participants with treatment-related Physical examination abnormality
  4. Number of participants with treatment-related Local response evaluation abnormality
  5. Number of participants with treatment-related Laboratory test abnormality
PK Characteristics of GV1001 | 2 weeks
  To evaluate the pharmacokinetic characteristics of GV1001 in healthy adults during both single and multiple administrations in different dose scheme.
  1. Part A: Cmax, AUClast, AUCinf, Tmax, t1/2, CL/F, Vz/F
  2. Part B, Extra cohort: Cmax, Cmax,ss, AUCτ, AUCτ,ss, Tmax, Tmax,ss, t1/2, t1/2,ss, CL/F, CLss/F, Vz/F, Vz,ss/F, Peak-trough fluctuation, Accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea